CLINICAL TRIAL: NCT05079698
Title: A Safety Study of Stereotactic Body Radiotherapy (SBRT) and 177Lu-PSMA617 for the Treatment of Hormone Sensitive, Oligometastatic Prostate Cancer
Brief Title: A Study of Stereotactic Body Radiotherapy and 177Lu-PSMA-617 for the Treatment of Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-158
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Stereotactic Body Radiotherapy; 177Lu-PSMA-617; 21-158
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; Radiosurgery

STUDY DESIGN:
Intervention Model Description: The study is a single-institutional pilot study of 6 total patients at MSKCC.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiotherapy and 177Lu-PSMA-617 (Experimental)
  Interventions: Drug: 177Lu-PSMA-617; Procedure: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Intravenous (IV) infusion of 177Lu-PSMA-617 on Day 1 of treatment Cycles 1 and 2. PSMA PET utilizing either the 68Ga-PSMA-11 or 18F-DCFPyL tracer is acceptable. Patients should be restaged using the same tracer which was utilized to establish initial eligibility for the trial.
Procedure: Stereotactic Body Radiotherapy (SBRT) — No later than 5 weeks (+/- 7 days) after the 2nd cycle of 177Lu-PSMA-617, patients will then undergo SBRT (900 cGy x 3 fractions).

SUMMARY:
The researchers are doing this study to find out whether giving 177Lu-PSMA-617 followed by a type of radiation therapy called SBRT (stereotactic body radiation therapy) is a safe treatment for your cancer. The study agent has been shown to target tumor cells, and the researchers think that adding 177Lu-PSMA-617 to SBRT may prevent or delay the cancer from continuing to spread.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have a biopsy proven adenocarcinoma of the prostate (biopsy confirmation of the primary tumor or oligometastatic tumor is acceptable)
* The patient's primary tumor must have been previously treated with surgery and/or definitive radiation. Prior salvage treatments (radiation or surgery) to the prostate bed or pelvis is allowed.
* Patients must have a negative multiparametric MRI and/or negative biopsy of the prostate (or prostate bed) even if other imaging modality (including PSMA) was negative for disease in the prostate (or prostate bed) within 2 months of enrollment on study

  °If patient is post-prostatectomy, the MRI Prostate can be excluded at clinician's discretion
* Patients must have had a PSMA scan within 2 months of enrollment on study
* Patient has not received any form of prostate-cancer directed therapy since undergoing screening PSMA scan
* Patient must have 1-5 oligometastatic tumors or lesions of the bone or soft tissue that are detectable on a PSMA PET scan.

  * Outside PSMA scans not performed at MSKCC are acceptable but will require official read by MSKCC nuclear medicine for confirmation of metastasis
  * Patients with sclerotic, non-PSMA avid osseous lesions which are not felt to reflect active metastatic disease by a radiologist are eligible for the protocol assuming they also have 1-5sites of PSMA avid disease as well as no non-PSMA avid sites which are felt to reflect active metastatic prostate cancer
* All oligometastatic lesions must be amenable to SBRT to a dose of 9 Gy x 3 without exceeding nationally recognized dose limits to adjacent organs at risk as deemed by the treating radiation oncologist
* Patient's insurance is willing to cover SBRT treatment or the patient agrees to cover the costs of this therapy
* Patient must have a prostate specific antigen (PSA) ≥ 0.2 ng/mL but ≤ 50 ng/mL
* Patient may have had prior systemic therapy and/or ADT associated with treatment of their primary prostate cancer. Patient may have had ADT associated with salvage radiation therapy.

  * Patients who have been on hormone therapy within 12 months of consent must have testosterone within normal range (221-716 ng/dL at MSKCC) in order to be eligible for treatment on study.
  * Baseline testosterone below the normal range for patients who have not had hormone therapy within 12 months of study entry is acceptable
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 or the equivalent KPS conversion value of ≥ 60 .
* Patient must have a serum creatinine level < 1.5 x ULN or EGFR > 60 mL/min
* Patient must have adequate liver laboratory values:

  * ALT and AST ≤ 2.5 x ULN
  * Albumin > 2 g/ dL
  * Bilirubin < 3 X ULN
* Patient must have normal organ and marrow function as defined as:

  * Total white blood count > 3.0 K/mcL
  * Absolute Neutrophil Count ≥ 1.5 K/mcL
  * Platelets ≥ 100 K/mcL
  * Hemoglobin ≥ 9 g/dL
* The effects of 177Lu-PSMA-617 and SBRT on the developing human fetus at the recommended therapeutic dose are unknown. Men (including men with vasectomies) must agree to use adequate contraception (a condom and another effective method of birth control) prior to registration, for the duration of study participation, and for at least 3 months thereafter. Men must also agree not to donate sperm for the duration of study participation, and for at least 3 months thereafter.
* Patient must be ≥ 18 years of age
* Ability to understand, and willingness to sign the informed consent

Exclusion Criteria:

* Pathological findings consistent with small cell and/or neuroendocrine carcinoma of the prostate or any other histology not consistent with prostate adenocarcinoma
* Patients with documented castration resistant prostate cancer (CRPC)
* Patients with a PSMA scan within 2 months of enrollment that do not demonstrate metastatic lesions or demonstrate more than 5 discrete metastatic lesions
* Patients with PSMA negative metastatic lesions or with a mixture of PSMA avid and PSMA negative disease
* Patients with metastatic lesions not amenable to SBRT or treatment of which using a 9 Gy x 3 regimen would result in exceeding nationally accepted or institutional dose limits for nearby organs at risk
* Patients with previous radiation therapy for oligometastatic disease are still eligible
* Patients with prior radiotherapy to > 25% of the skeleton or prior exposure to prior 223Radium, 89Strontium or 153Samarium containing compounds
* Patients with spinal cord compression, impending spinal cord compression, or parenchymal brain metastases (patients with epidural disease without cord compression are eligible)
* History of a prior or concurrent malignancy whose natural history or treatment has potential to interfere with the safety or efficacy assessments
* Patients with known or suspected history of grade II or higher chronic kidney disease (CKD)
* Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to registration.
* Seizure or known condition that may predispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to enrollment, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
* Gastrointestinal disorder affecting absorption
* History of viral hepatitis or chronic liver disease with active symptoms
* History of pituitary or adrenal dysfunction
* Previously diagnosed active infection (e.g., human immunodeficiency virus [HIV] or viral hepatitis)
* Any condition that in the opinion of the investigator, would preclude participation in this study
* Concurrent corticosteroids and/or adrenal hormone inhibitors, PC-SPES, finasteride, or dutasteride is not allowed.
* Receipt of any other investigational agents or participation in a concurrent treatment protocol
* Inability to life flat during or tolerate PET CT/MR or SBRT
* Patients must not have claustrophobia that would preclude PET/CT imaging or other contraindications to CT imaging
* Known allergies, hypersensitivities, or intolerance to Lu-PSMA-617 or its inactive compounding components

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 27 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with dose limiting toxicity (DLT) of fractionated dose of 177Lu-PSMA-617 (Pilot) | 1 year
  using the National Cancer Institute CTCAE, Version 5

SECONDARY OUTCOMES:
Proportion of subjects with dose limiting toxicity (DLT) of fractionated dose of 177Lu-PSMA-617 (Phase I) | 1 year
  National Cancer Institute CTCAE, Version 5 will be used for determining the severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Imber, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm